CLINICAL TRIAL: NCT00955188
Title: Evaluating a Preference-tailored Intervention to Increase CRC Screening in Primary Care Settings
Brief Title: Computer-Based Tailored or Standard Information for Colorectal Cancer Screening
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000632080; R01CA131041 (NIH); P30CA046592 (NIH); H8000-32900-01
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: computer-assisted intervention
Other: educational intervention
Other: medical chart review

SUMMARY:
RATIONALE: A computer program that provides information on colorectal cancer screening based on a patient's test preferences may be more effective than a computer program that gives standard information in helping patients get regular colorectal cancer screenings.

PURPOSE: This randomized clinical trial is studying computer-based tailored information to see how well it works compared with standard information for colorectal cancer screening.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the effectiveness of a preference-tailored (PT) intervention vs standard information (SI) delivered via computer for increasing patients' adherence to colorectal cancer (CRC)-screening guidelines in a randomized controlled trial in two racially/ethnically diverse geographic locations.
* To assess the impact of the intervention on patient perceptions of informed-decision making, physician recommendation for CRC screening, decision conflict and satisfaction, and intention to get screened 3 days after a primary care visit.
* To conduct a cost-effectiveness analysis of a preference-tailored strategy for increasing CRC screening utilization.

OUTLINE: This is a multicenter study. Patients are randomized by the computer program to 1 of 3 intervention arms.

* Arm I (preference-tailored intervention): Patients receive overview information about colorectal cancer (CRC), including graphics and descriptions of the colon and colon polyps. Patients then complete a preference-assessment exercise test by using a specially designed website. A brief description of the test is given at this time, and patients are offered the option to learn more about their preference-matched test. Patients are then given a list of other available CRC-screening tests with a brief description and option to learn more about each test. The program informs them when all information has been viewed. At the time the patients exit the program, or have viewed all the information available, they are asked to choose which test is preferable to receive from a list of existing test options.
* Arm II (standard information intervention): Patients receive overview information as in arm I. The patients then use a website listing of the four existing CRC screening test options along with graphical representations. They are allowed to interact with this web page to view basic or more information about any or all of the tests. The program informs them when all the information has been viewed. At this point, patients are asked to choose which test they would prefer to receive from a list of existing test options, as in arm I.
* Arm III (usual care): Patients receive usual care and do not receive any extra educational materials. Patients may receive a telephone follow up at 12 months.

Upon completion of the intervention, patients in arms I and II receive a printout to take with them to their upcoming appointment. For those in arm I, this printout will include their top three attributes, their preference-matched test, and their final test choice. For those in arm II, this printout will include a list of the four screening tests but will not list their final test choice.

Patients in arm I and II undergo a 3-day follow-up telephone interview. Medical charts of all patients in all 3 arms are reviewed at 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At average risk for colorectal cancer (CRC), defined as the following:

  * No personal history of CRC, adenomatous colon polyps, or inflammatory bowel disease
  * No family history of CRC
* Not up-to-date with CRC screening in past year OR have never been screened, defined as

  * Up-to-date screening is defined as having completed 1 of the following:

    * Fecal occult blood test within the past 2 years
    * Sigmoidoscopy within the past 5 years
    * Colonoscopy with the past 10 years
    * Double-contrast barium enema within the past 5 years
* Patient at San Francisco Community Health Network or at Henry Ford Health System and a member of the Health Alliance Plan

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 1 year
* No history of inflammatory bowel disease, polyposis, or hereditary nonpolyposis
* No severe comorbidity or significantly lowered life expectancy, including any of the following:

  * Do not resuscitate (DNR)/do not intubate (DNI) code status
  * Metastatic cancer
  * End-stage congestive heart failure
  * Severe chronic obstructive pulmonary disease
  * Coronary artery disease with recent myocardial infarction or unstable angina
  * Dementia

PRIOR CONCURRENT THERAPY:

* No prior bowel resection

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kelsey-Seybold Clinic, Houston, Tx
  Study Coordinator: Bettencourt , Judy ( ) Email: Judith.L.Bettencourt@uth.tmc.e Phone: 713-500-9754
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2004-08; Primary Completion 2007-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Adherence to colorectal cancer screening at 12 months post-intervention | 12 months

SECONDARY OUTCOMES:
Elements of informed decision making | 12 months
Knowledge about screening options | 12 months
Decisional conflict and satisfaction | 12 months
Intention to get screened | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah T. Hawley, PhD, MPH, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan